CLINICAL TRIAL: NCT06689293
Title: Faecal Immunochemical Tests (FIT) for Surveillance After Colorectal Cancer (CRC) Study
Acronym: FITS
Status: Recruiting | Type: Observational
Sponsor: Nottingham University Hospitals NHS Trust (Other)
Responsible Party: Sponsor
Other Study IDs: 22CR002
Record Dates: First submitted 2024-11-12; First posted 2024-11-14 (Actual); Last update posted 2026-01-21 (Actual); Status verified 2026-01

CONDITIONS: Colorectal Cancer (CRC)
Keywords: colorectal; Faecal Immunochemical Testing (FIT); surveillance
MeSH Terms: conditions — Colorectal Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Study group: Participants aged over 18 with previous colorectal cancer resection for curative intent, excluding those with current ileostomy or recurrent cancer.
  Interventions: Diagnostic Test: Faecal Immunochemical Test

INTERVENTIONS:
Diagnostic Test: Faecal Immunochemical Test — Self-collected sample from stool collected into testing kit

SUMMARY:
In the United Kingdom, over 25,000 patients have an operation for bowel cancer each year. After their operation, patients are monitored with a colonoscopy (camera test of the bowel) approximately 3 years after their operation, to look for any possible return of the cancer. Colonoscopies, and the bowel-cleaning medications needed, can be unpleasant for patients.

The Faecal Immunochemical Test (FIT) is a test to look for blood hidden in the poo. Blood in the poo can be a sign of bowel cancer, or a growth that can turn in to a cancer if left untreated (polyps). We currently use this test for bowel cancer screening, and to assess the risk of cancer in patients with bowel symptoms. You may have had a FIT when having tests for bowel cancer. We know this test is effective in picking up bowel cancer in these cases, but its use has not been assessed in following-up patients who have had treatment for bowel cancer previously.

For this study, we aim to see if a FIT stool sample test is accurate at diagnosing a return of bowel cancer for patients who have had a previous operation for bowel cancer. We want to see if using FIT could 'rule-out' cancer for some patients and be a potential alternative to colonoscopy for some patients in the future, allowing them to avoid this sometimes unpleasant test, which patient groups have told us is important for them.

Patients taking part in this study will have their usual treatment, including their colonoscopy (or sometimes a scan of the bowel), but will be asked to also provide a single FIT sample to assess how accurate this test is. The FIT sample is a quick and easy test of the poo that you can take at home and send to Nottingham University Hospitals NHS Trust (NUH) for testing. It should take no more than 5 to 10 minutes to take the sample, and a prepaid envelope is included to send the sample back to NUH for testing.

We aim to include at least 1,000 patients across 7 hospital trusts in the East Midlands.

DETAILED DESCRIPTION:
This is a diagnostic accuracy study, to assess the accuracy of FIT for predicting recurrence of CRC, or other significant pathology such as polyps and Inflammatory Bowel Disease (IBD), for patients undergoing their 3-year surveillance colonoscopy/CT Colon (CTC). Patients will be recruited from across 7 Hospital Trusts in the East Midlands. Eligible patients will be those adult patients who have had a curative operation for bowel cancer, due their surveillance colonoscopy/CTC. Patients with their entire colon removed, or with current ileostomy, will be excluded. The target would be for the patient to be recruited and complete their sample within the 3 months prior to the colonoscopy or CTC.

Eligible patients will be identified at each site and sent a postal study pack including Patient Information Sheet (PIS), consent form and FIT sampling kit. Patients agreeing to take part need only return the sample and consent form. They will go on to receive their normal care (surveillance colonoscopy or CTC), with the patients and clinicians responsible for their surveillance being blinded to the FIT result. The FIT samples will be analysed in NUH, and the results compared to the outcomes of the surveillance colonoscopies (or CTC) performed at the local Trusts. This will be used to see how accurate FIT is at predicting CRC recurrence, significant polyps and IBD. Patients will have no change to their normal care.

RESEARCH QUESTION / AIM(S) To assess how accurate a simple poo test (FIT) is in diagnosing bowel cancers and polyps (growths in the wall of the bowel) at high-risk of turning in to a cancer in patients who have had an operation for bowel cancer in the past.

Objectives

The primary objective is to assess the accuracy of FIT for recurrent colorectal cancer or high-risk polyps (high risk for turning in to a cancer if untreated) in patients having their 3-year surveillance colonoscopy/CTC after previous curative operation.

The secondary objective is to assess the accuracy of FIT for lower-risk polyps and inflammatory bowel disease in these same patients. We will also assess whether any demographic differences in the patients affect FIT-return rate.

Outcome To measure the diagnostic accuracy of FIT for the primary and secondary objectives above, compared with the reference of surveillance colonoscopy/CTC 3 years after bowel cancer surgery, in terms of sensitivity, specificity, positive predictive value and negative predictive value. For CRC and significant polyps, we will also generate a 'Number Needed to Scope' (NNS) for various FIT thresholds.

STUDY DESIGN AND METHODS OF DATA/SAMPLE COLLECTION AND DATA/SAMPLE ANALYSIS Patients who have had an operation for bowel cancer are invited for a colonoscopy (camera test of the bowel) or CTC (a special type of scan of the bowel) approximately three years after their operation to look for any potential return of the cancer within the bowel. All adult patients due to have their colonoscopy/CTC after having had an operation for bowel cancer three years prior across the East Midlands will be invited to the study. The only patients that will be excluded are those with a certain type of stoma present made from the small bowel (ileostomy), as these patients do not pass faeces from the large bowel.

Each hospital in the region has a computer database for when patients are due their surveillance colonoscopy/CTC after previous operation for bowel cancer. All hospitals in the region have agreed to take part in the study, including: Nottingham University Hospitals (NUH), Royal Derby Hospital, Chesterfield Royal Hospital Foundation Trust, Sherwood Forest Hospitals NHS Foundation Trust , United Lincolnshire Hospitals Trust, University Hospitals of Leicester NHS Trust and Northampton General Hospital NHS Trust. The study will be run from NUH, with day-to-day running of the study overseen by a research fellow and Associate Professor of Surgery. A wide-range of hospitals ensures we can include a diverse range of patients from many different ethnicities and backgrounds.

Clinical teams at each Trust will identify a list of patients to invite to the study. Sites will send out information about the study to eligible patients. Packs sent to the patients by sites will include a letter explaining the study, a Patient Information Leaflet, a consent form to sign if they consent to the study (including for the transfer of information to NUH), a FIT-sample return kit with prepaid stamp-addressed return envelope and contact details for the research team should they wish to discuss the study further. The FIT-sample kit, and all study documents, will be dispatched from packs held by each hospital site and returned to the testing laboratory at NUH.

Patients choosing to participate in the study will receive their normal care, including having their colonoscopy/CTC as planned. The only difference is that they will be asked to send a FIT sample to us (the research team at NUH), at no cost to the patient, ideally within the 3 months prior to their surveillance colonoscopy or CTC. The FIT result will not be revealed to the patient or clinical team, to remove any risk that it may impact the clinical care of the patient. Therefore, the only difference for the patient in participating in the study is providing the FIT sample, as their clinical care will not be affected by the study. This is clearly described in the Patient Information Leaflet. This means patients, clinicians and outcome assessors (who review clinical outcomes of colonoscopies/CTCs at each site) will be blinded to the FIT result so it cannot impact care or results.

We expect a high response rate. Previous studies in Nottingham have shown >90% of patients respond to a postal request for a FIT, understanding the role it has in detecting cancer. Almost all patients accept a colonoscopy, being familiar with its role in detecting their initial cancer. In Nottingham, less than 5% of patients refuse their colonoscopy 3 years after cancer surgery. For these patients, a scan of their tummy (CT colonoscopy (CTC)) will be offered instead, and these patients will still be eligible for inclusion in this study if they have received this test. The research team at each site will review the results of the colonoscopy or scan and upload this to a secure, anonymised online portal for data entry, along with information on the operations performed, clinical outcomes for the patient and details on the most recent blood tests such as CEA, haemoglobin level and platelets.

FIT results for patients will be compared with their findings from their colonoscopy or CTC. We will see if a high result is related to the risk a patient had a bowel cancer found, or if a low result is effective to "rule-out" cancer. The same tests will be done to see how effective FIT is for high-risk polyps, low-risk polyps and inflammatory conditions of the bowel.

We estimate we need 1,000 patients to join the study to be able to show an effect. Data from all the hospitals shows that we have approximately 1,050 patients who are eligible per year. We will run the study for 18 months, expecting around 1,575 eligible patients in this time. This requires less than two-thirds (63% of patients) to respond to the study, which is much less than what we have seen in previous studies. If required, we will be able to run the study to 24 months if recruitment is insufficient.

All data analysis will be done at NUH and the university of Nottingham. Prior to data being sent to the UoN for analysis, the data will be re-coded, and only the central team at NUH, will hold this subsequent pseudonymisation key.

The details of those patients approached will be logged at each local hospital site, using a screening log. Patients returning a sample and consent form will be logged by the NUH lab in an enrolment log on the Colorectal Research drive at NUH (in a folder than can only be accessed by the researchers). The study sites will then be informed of those who have returned the consent and sample and a copy of the consent forms will be sent to the relevant local sites, to enable sites to create REDCap entries for collection of the study data. Transfer of the enrolment log of patients who have consented to involvement, and relevant consent forms, from NUH to the relevant site will be via secure, encrypted email (NHSmail). Research teams at each study site will upload pseudonymised information securely to REDCap detailing the outcomes of colonoscopy/CTC, as well as demographic information and details of their initial operation. The REDCap IDs of these pseudonymised entries will be linked to patient FIT samples to allow matching of the FIT results at NUH to patient outcomes. All identifiable patient information will be secured either on password-protected electronic files on the NHS network at each hospital, or within the study folder kept in a locked room (each study site having a list of their own patients linked to REDCap IDs, the research team at NUH having a list of all patients recruited (study ID number and name only, with FIT result) so FIT samples can be linked to patients to allow analysis of outcomes).

Only the research team at NUH will have access to the FIT results, so the results cannot be used to influence patient care. Each site will only have access to information for their own hospital trust. FIT samples will all be analysed at the NUH Bowel Cancer Screening Programme laboratory and disposed of when analysis is complete.

Statistical analysis will be done using R.

STUDY SETTING This is a multicentre study running across 7 hospital trusts in the East Midlands. Each participating site has their own database for which patients are due their 3-year surveillance colonoscopy or CTC. Each site will have a number of premade study packs with unique Study ID, allowing each site to recruit patients by posting of study packs including PIS, consent forms and FIT sampling kits. This will clearly explain the study and how to take the FIT sample. All sequential patients in the study period will be assessed for eligibility and recruitment. Patients will be recruited from a multitude of sites to allow the numbers and power to look for a relatively rare outcome of recurrent CRC. The entire East Midlands is included, so that the results are representative of the region as a whole.

All analysis of FIT samples regionally currently takes place at NUH. Therefore, our laboratory is best-placed for the analysis of returned samples. This also allows the blinding of clinicians at each site to the FIT result so it cannot impact treatment; only the research team (who have no care responsibilities for the patients) will be able to access the results. Teams at participating sites are responsible for highlighting eligible patients and sending out the packs for recruitment, then following up the outcomes of those participating to upload onto REDCap. NUH will have access to the FIT result for each study ID, as well as the details uploaded for each study ID on REDCap.

As clinical outcomes of colonoscopy/CTC are only available at each site, research teams employed by each participating trust will collect the outcomes for the study and upload this in pseudo-anonymous format to REDCap. The REDCap ID (the same as Study ID) will be linked to patient identifiers in the site files, to maintain confidentiality but allow linkage of FIT results to clinical outcomes. Oversight of the study at each site will be managed by a PI at each site who is a practising clinician there, with the CI for the study based within the research team at NUH.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years
* Histological diagnosis of colorectal carcinoma
* Previously treated by surgical resection with curative intent for colorectal carcinoma
* Due whole-colon investigation for CRC follow-up as part of local routine care (Colonoscopy or CT colon)

Exclusion Criteria:

* Patients under the age of 18
* Patients unable to give valid informed consent
* Patients with a current ileostomy, or no remaining colon after their operation (patients with colostomy will not be excluded)
* Patients already diagnosed with recurrence of their colorectal cancer

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Eligible patients, due to have their 3-year postoperative surveillance colonoscopy/CTC, at each site will be invited to participate in the study. The colorectal cancer lead in each Trust has agreed to support the study and actively recruit from their site.
  Patients will be identified at each site by the clinical teams based there. Each trust has a locally managed electronic database used to manage surveillance scheduling of investigations for patients following CRC surgery. Participating Trusts include Nottingham University Hospitals [NUH], Royal Derby Hospitals [RDH], Chesterfield Royal Hospital Foundation Trust [CRHFT], Sherwood Forest Hospitals NHS Foundation Trust [SFHFT], United Lincolnshire Hospitals Trust [ULHT], University Hospitals of Leicester NHS Trust [UHLT] and Northampton General Hospital NHS Trust [NGHT].
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2025-02-28 (Actual); Primary Completion 2027-02 (Estimated); Study Completion 2027-06-23 (Estimated)

PRIMARY OUTCOMES:
Recurrent colorectal cancer or high-risk polyps | Surveillance colonoscopy within 3 months of FIT sample
  Presence of colorectal cancer (recurrent) or high-risk polyp (>10mm, high-grade dysplasia) at 3-year surveillance colonoscopy or CT colon

SECONDARY OUTCOMES:
Low-risk polyps or inflammatory bowel disease | Surveillance colonoscopy within 3 months of FIT sample
  Low -risk (<10mm) polyps or inflammatory bowel disease found at surveillance colonoscopy or CT colon.
Demographics of those not returning a FIT prior to surveillance colonoscopy | Surveillance colonoscopy within 3 months of FIT sample
  Age, sex, ethnicity and deprivation level (from first 4 characters of post code) compared between those returning and not returning a FIT.

CONTACTS AND LOCATIONS:
Locations (1):
- Nottingham University Hospitals NHS Trust, Nottingham, United Kingdom